CLINICAL TRIAL: NCT07143084
Title: Investigation of the Relationship Between Nutritional Status Assessment and Frailty in Critical Care Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayşe EKEN, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: 02.05.2025_E-25-426
Record Dates: First submitted 2025-06-25; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-05

CONDITIONS: Fraility; Critical Illness
Keywords: CONUT; Fraility; NUTRIC Score
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Patients above 65 years old

SUMMARY:
This study aims to understand the effects of these two parameters on clinical outcomes by examining the relationship between NUTRIC and CONUT scores in intensive care patients. The results of the study may contribute to the development of new approaches to the treatment process of patients by better understanding the relationship between nutritional status and pre-hospital frailty in intensive care units. In addition, eliminating the deficiencies in this area will pave the way for the creation of more effective and personalized treatment plans for similar patients.

ELIGIBILITY:
Inclusion Criteria:

* over 65
* 48 hours min. ICU stay

Exclusion Criteria:

* Patients who are under 65 years of age
* whose intensive care stay does not exceed 48 hours
* who have missing data for serum albumin or lymphocyte count or total cholesterol,
* who have been diagnosed with hematological diseases such as leukemia or lymphoma

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Over 65 years, critically ill patients, who are submitted to ICU.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between CONUT scale and frailty in intensive care patients | From enrollment 2 days
  To evaluate the correlation between the CONUT scale and frailty, Pearson or Spearman correlation analysis will be performed depending on suitability for normal distribution. Logistic regression analysis will be performed to assess the independent association between CONUT scale and frailty. Potential confounding variables such as age, gender, APACHE II score, and activities of daily living will be included in the regression model.

SECONDARY OUTCOMES:
Association of NUTRIC score and CONUT scale with clinical outcomes | From enrollment to through study completion an average of 1 year
  To evaluate the correlation between the NUTRIC score and CONUT scale with clinical outcome, Pearson or Spearman correlation analysis will be performed depending on suitability for normal distribution. Logistic regression analysis will be performed to assess the independent association between CONUT scale and NUTRIC score. Potential confounding variables such as age, gender, APACHE II score, and activities of daily living will be included in the regression model.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training And Research Hospital, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Auza-Santivañez, J. C., Perez, J. S., Lara, Y. D., León, D. O., Condori-Villca, N., & Loaces, J. P. A. Predictive value of the CONUT scale in the early detection of nutritional risk and its relationship with mortality in critically ill patients.
- [Background] Kos, M., Titiz, H., Onec, B., Soysal, T., Kutlucan, A., Emen, S. S., & Kutlucan, L. (2016). Association of "controlling nutritional status index" and "prognostic nutritional index" with intensive care unit survival in elderly patients. European Geriatric Medicine, 7(1), 13-17.
- [Background] Lo Buglio A, Bellanti F, Capurso C, Vendemiale G. Controlling Nutritional Status (CONUT) Score as a Predictive Marker in Hospitalized Frail Elderly Patients. J Pers Med. 2023 Jul 10;13(7):1119. doi: 10.3390/jpm13071119. PMID 37511732